CLINICAL TRIAL: NCT02225379
Title: Development and Assessment of Feasibility of Non-invasive Multiple Sensor Hypo-Sense Sensor as a Tool for Detection of Hypoglycemia - Exploratory Study for Prototype Rev 1
Brief Title: Development and Assessment of Feasibility of Non-invasive Multiple Sensor Hypo-Sense as a Tool for Detection of Hypoglycemia
Acronym: Hypo-Sense
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Collaborators: Night Sense Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 029514ctil
Record Dates: First submitted 2014-07-29; First posted 2014-08-26 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Type 1 Diabetes; Nocturnal Hypoglycemia
Keywords: Type 1 Diabetes; Hypoglycemia detection; Non-invasive sensor; Nocturnal hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypo-Sense (non invasive sensor) (Experimental): Parallel measurements of capillary blood glucose using reference method and data generated by the non- invasive study device (Hypo Sense) during approximately 4 hours, in which a hypoglycemic event will be induced.
  Interventions: Device: Hypo-Sense (non invasive sensor)

INTERVENTIONS:
Device: Hypo-Sense (non invasive sensor) — Parallel measurements of capillary blood glucose using reference methods (both capillary glucometer and continuous sensor) and data generated by the non- invasive study device during approximately 4 hours, in which a hypoglycemic event will be induced.

SUMMARY:
Hypo Sense is a non- invasive method for detection of hypoglycemia. The Hypo Sense combines an array of non-invasive sensors which monitors the patient's physiological parameters (heart & respiration rate, perspiration, skin temperature and arm motion) designed as a wrist watch device.

The Hypo sense is intended for monitoring symptoms of hypoglycemia in diabetic patients in hospital environment among type 1 and type 2 diabetes adults as an adjunctive device to reference methods

The proposed study will be consisting of two main segments:

The primary aim of segment 1 of the study is data collection and calibration of the Hypo Sense sensor prototype compared to standard invasive reference glucometer.

The primary aim of segment 2 of the study is to validate the Hypo Sense prototype performance in detecting hypoglycemic events.

During the first segment of the study we intend to collect in parallel measurements of blood glucose using reference method (capillary glucometer) and continuous data generated by the non- invasive study device during approximately 4 hours, in which a hypoglycemic event will be induced.

The reference and study device data will be analyzed using multivariate regression model to formulate a calibration algorithm model. This model will translate the set of the physiological recorded parameters into detection of hypoglycemic events.

During the second segment of the study we intend to evaluate the validity of the Hypo Sense sensor ability to detect hypoglycemic events compared to standard invasive reference method (capillary glucometer).

ELIGIBILITY:
Inclusion Criteria:

* Signing an inform consent form prior to any trial related procedure
* Type 1 diabetes diagnosed at least 12 months prior to study inclusion
* Age > 18 years old

Exclusion Criteria:

* Participating in other device or drug study
* Any significant disease or condition, including psychiatric disorders that in the opinion of the investigator is likely to affect patient's compliance or ability to complete the study
* Patients with one or more of the following diseases: malignancy, myocardial insufficiency, nephrologic disease or any other chronic disease
* Chronic skin problem in the lower inner arm
* Pregnant or breast feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Sensitivity | At final visit ( week 4 for participants at segment 1 of the study and week 6 for participants at segment 2 of the study)
  Sensitivity of the Hypo Sense-the proportion of hypoglycemia events detected by the Hypo Sense sensor from total number of hypoglycemic events detected by reference capillary glucometer
Positive Predictive Value of the hypo-Sense | At final visit ( week 4 for participants at segment 1 of the study and week 6 for participants at segment 2 of the study)
  Positive Predictive Value of the hypo sense- the proportion of validated ("true") hypoglycemia events detected by the hypo sense sensor from total alerts detected by the Hypo-Sense sensor

CONTACTS AND LOCATIONS:
Overall Officials: M Phillip, Prof, Principal Investigator — Schneider Children's Medical Center
Locations (1):
- Schneider Children's Medical Center, Petah Tikva, Israel